| 1 | Violet Light for the Treatment of Myopia |
|---|---|
| 2 | |
| 3 | Version 6.0 |
| 4 | July 2, 2023 |
| 5 | |
| 6 | |
| 7 | Principal Investigator: Melissa Rice, OD |
| 8 | <b>Sub-Investigators:</b> Richard Lang, PhD, Veeral Shah, MD, PhD, Kelsey Carriere, OD, Katherine Hogan, OD, Kelsey Mach, OD, Kelly Hayden, OD |
| 10 | Virginia Utz, MD, Anne Slavotinek, MD |
| 11 | |
| 12 | |
| 13 | |
| 14 | |
| 15 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 20 | |
| 21 | |
| 22 | |

#### **Table of Contents** 24 25 1. Background and Summary 26 1.1 Epidemiology and Disease Burden 27 1.2 Current Treatments 28 1.3 Myopia and Violet Light 29 1.4 Role of Genetics in Myopia 30 1.5 Bios SkyView Lamps 31 1.6 Impact of UV Blocking Lenses 32 1.7 Study Design 33 1.7 (A) Study Groups 34 1.7 (B) Designating Dawn and Dusk 35 1.7 (C) Onset HOBO Occupancy Sensor (UX90-005M) 36 1.7 (D) DNA Storage via Saliva 37 1.8 Study Objective 38 1.9 Timing of Intervention and Outcome for Proposed Study 39 2. Considerations 40 2.1 Risks 41 2.2 Risk of Examination Procedures 42 2.3 Risk Assessment 43 2.4 Reporting of Adverse Events 44 2.5 Study Costs 3. Study Outline 45 46 4. Enrollment 47 4.1 Eligibility Assessment 48 4.2 Inclusion Criteria 49 4.3 Exclusion Criteria 50 4.4 Sample Size 51 4.5 Historical Information 52 4.6 Survey to Determine Lighting Schedule 53 4.7 Testing at the Enrollment Visit 54 4.8 Refractive Correction 55 5. Randomization 56 **5.1 Randomization Process** 57 6. Equipment Pickup Visit 58 6.1 Prescription Glasses 59 6.2 Study Lamp 60 6.3 HOBO Sensor 61 6.4 Automated Wall Plug-In 62 6.5 Testing Not Completed at Enrollment 63 7. Follow-Up 64 7.1 REDCap Daily Surveys 65 7.2 Telephone Calls 66 7.3 Follow-Up Visits: 6-Month and 12-Month 67 7.4 Management of Refractive Error 68 7.5 Non-Randomized Treatment Other than Refractive Correction 69 7.6 General Considerations 70

8. Miscellaneous Considerations

8.1 Participant Withdrawals

71

| 72 | 8.2 Discontinuation of Study |
|---|---|
| 73<br>74 | <ul><li>8.3 Payment to Participants</li><li>8.4 Costs Covered by the Study</li></ul> |
| 7 <del>4</del><br>75 | 8.5 Costs Not Covered by the Study |
| 76 | 9. Data Storage and Analysis |
| 77 | 9.1 Analysis |
| 78 | 9.2 Decision Guideline |
| 79 | 9.3 Data Safety Monitoring Plan |
| 80 | 9.4 Source Documents and Case Report Forms |
| 81 | 9.5 Changes to Protocol |
| 82 | 10. References |
| 83 | |
| 84 | |
| 85 | |
| 86 | |
| 87 | |
| 88 | |
| 89 | |
| 90 | |
| 91 | |
| 92 | |
| 93 | |
| 94 | |
| 95 | |
| 96 | |
| 97 | |
| 98 | |
| 99 | |
| 100 | |
| 101 | |

103

104

118

# 1. Background and Summary

### 1.1 Epidemiology and Disease Burden

- Myopia (shortsightedness) is the most common eye condition in the world and is only increasing in
- prevalence, with studies predicting 4.7 billion afflicted by 2050. This increase in prevalence is
- particularly notable in East Asia, but myopia is increasing in the US as well: a study done with a
- 108 contemporary American cohort in Southern California found that 41.9% of the cohort, aged 5-19 years
- old, were myopic.<sup>2,3</sup> Although visual impairment caused by myopia is generally correctable (via glasses,
- contact lenses, etc.), uncorrected refractive error costs \$202 billion annually in global GDP.<sup>2,3</sup> High
- myopia is associated with increased risks of glaucoma, cataracts, and retinal detachment.<sup>4-6</sup>

### 112 1.2 Current Treatments

- 113 Slowing the progression of myopia has been attempted through a range of treatments with varying
- degrees of success. Among the most promising have been soft bifocal contact lenses, orthokeratology,
- and antimuscarinic agents (pirenzepine, atropine, etc.). <sup>7,8</sup> However, these treatments are not without
- side effects: atropine can cause side effects such as photophobia, and orthokeratology carries the risk of
- microbial keratosis. 9 In addition, compliance with contact lens wear can be poor. 10

### 1.3 Myopia and Violet Light

- An abundance of studies have shown that outdoors exposure is protective against myopia onset. 11-16
- Meta-analysis indicates that one additional hour spent outdoors per week translated to a 2% reduced
- odds of developing myopia. 14 Some studies have also shown that outdoor exposure can reduce myopic
- progression. 14,16 The mechanism for this is yet unclear, but it has been theorized that violet light may be
- 123 key to this protective effect. 17 Due to overzealous UV protection, violet wavelengths have been rendered
- nearly absent from modern life despite being part of the visible spectrum: windows have very low
- transmittance for wavelengths below 400 nm, indoor lighting does not incorporate violet, and UV
- 126 blocking glasses and contact lenses are abundant. 17
- 127 Previous studies by Torii et al. indicated that violet light is protective against myopia progression in
- humans. A retrospective study compared patients wearing non-violet transmitting eyeglasses, partially
- violet-blocking contact lenses, and violet light transmitting contact lenses, and found that patients
- 130 wearing violet light transmitting contact lenses had a significantly decreased amount of myopia
- progression as measured by axial length elongation. <sup>17</sup> Additionally, violet light was shown to influence
- 132 high adult myopia: patients who received non violet light transmitting phakic intraocular lens
- implantations were significantly more myopic than patients who received violet light transmitting
- 134 implantations.<sup>18</sup>
- Animal studies indicate that the light-sensitive protein OPN5 may be key in violet-light mediated
- 136 suppression of myopia. OPN5 has previously been shown to regulate light-dependent vascular
- development in the murine eye via suppression of vitreal dopamine, which simultaneously increased
- 138 retinal dopamine. 19 This is significant because retinal dopamine has been widely hypothesized to
- antagonize myopia development.<sup>20,21</sup> Violet light has been shown to reduce axial length elongation in
- 140 chicks as well as stimulate a higher long-term retinal dopamine level than blue, red, or white light. 17,21

141 Most recently, OPN5 has been shown to be necessary for violet-light mediated suppression of lens 142 defocus-induced myopia in mice. Violet light delivered for 3 hours in the evening (pre-dusk) protected 143 mice from lens defocus-induced myopia, an effect that was shown to be both time and wavelength 144 dependent – but did not protect OPN5 conditional null mice.<sup>22</sup>

### 1.4 Role of Genetics in Myopia

- Large-scale genetic studies have been performed in myopia and have implicated the important role of genetic factors. Through molecular techniques, such as linkage analysis, association studies, and sequencing analysis, many of the genes associated with myopia have been identified.<sup>23</sup> Furthermore, the prevalence of myopia increases significantly with the number of myopic parents; the associated development risk rates are 7.6% for no myopic parents, 14.9% for one myopic parent, and 43.6% for two myopic parents.<sup>24</sup> The evidence is conclusive of a genetic contribution to myopia beyond environmental factors, and exploring the genetic component of patients with myopia is critical in better understanding
- the disease.

145

154

163

170

171

174

175

176

177

178

### 1.5 Bios SkyView Lamps

- 155 In order to effectively deliver violet light, the BIOS SkyView lamp will be used. BIOS lighting uses
- patented circadian lighting technology to produce the highest melanopic to photopic lux ratio for a given
- 157 color temperature, translating to better equivalent melanopic lux for a lower correlated color
- temperature than other LEDs.<sup>25</sup> The BIOS SkyView lamps are equipped with wavelength-specific LEDs,
- able to provide a full profile of violet light (385 nm) for the purpose of this study.<sup>26</sup> The SkyView lamps
- have been approved by CCHMC for research use (assessment ID: 109744). The Aooshine bedside lamps,
- which will act as the control light source, have also been approved by CCHMC for research use
- 162 (assessment ID: 133975).

### 1.6 Impact of UV Blocking Lenses

- 164 UV blocking glasses are ubiquitous in modern society. Pediatric patients are commonly prescribed
- polycarbonate eyeglasses due to their innate UV-blocking capabilities and shatter resistance.<sup>25</sup> However,
- polycarbonate also attenuates the violet wavelengths that could potentially be crucial to myopia
- 167 control. 17,18,22 UV-blocking glasses, which typically seek to block wavelengths below 400 nm in an
- overabundance of caution, result in the elimination of much of the violet spectrum (380 nm to 450 nm),
- and could potentially be a contributing factor to the myopia epidemic.

### 4.9 Study Design

### A) Study Groups:

- To assess the effects of violet light and potential contribution from UV-blocking glasses, three study groups will be established:
  - A group (n = 24) will use the BIOS SkyView lamp with violet LEDs enabled for at least one hour during dawn and at least one hour during dusk. The group will wear CR-39 (UV-transmitting).
    - 2. A group (n = 24) will use the BIOS SkyView lamp with violet LEDs enabled for at least one hour during dawn and at least one hour during dusk. The group will wear polycarbonate (UV-blocking) glasses for the duration of the study.

3. A group (n = 24) will use the Aooshine lamp without any violet LEDs enabled for at least one hour during dawn and at least one hour during dusk. The group will wear CR-39 (UVtransmitting).

The study lamp (BIOS or Aooshine) should be the sole source of artificial illumination in participant rooms for the duration of lamp exposure, and throughout the study, exposure to natural light during designated dawn and dusk times should be minimized. Light is a noninvasive source of therapy, and as such, tracking the actual exposure to the lamps and compliance to the study design can be difficult. Therefore, the HOBO Occupancy Sensor (UX90-005), which measures movements of heat emitted by people in motion via passive infrared technology, will be paired with each BIOS lamp.

### B) Designating Dawn and Dusk

The best times for the SkyView and Aooshine lamps to undergo the dawn and dusk transition will be chosen individually per participant based on their anticipated daily schedule to maximize effectiveness. Each participant will be given a survey prior to enrollment so that research staff can determine the optimal times on an individual basis.

The one-hour timeframe is chosen to be consistent with known biological responses and the length of the natural dawn/dusk transition. The SkyView/Aooshine lamp will automatically turn on at dawn and automatically turn off after dusk. Both dawn and dusk are chosen because while dusk exposure was protective in the murine myopia model, this effect may be present at dawn in diurnal mammals.<sup>22</sup>

### C) Onset HOBO Occupancy Sensor (UX90-005M)

As light is a noninvasive form of treatment, assessing the amount of 'light' received is difficult to quantify in measuring the efficacy of violet light in slowing the progression of myopia. The Onset HOBO Occupancy Sensor uses infrared technology to measure fluctuations of temperature within a 5-meter radius. The temperature fluctuation readings are logged as numerical data which can then be retrospectively collected to then measure exposure to light during the duration of the study.

### D) DNA Storage via Saliva

In addition to exploring the efficacy of violet light exposure in treating myopia, the effects of genetic factors will be assessed from DNA extraction for research purposes only. In recent years, alongside the advent of more sophisticated molecular techniques such as linkage analysis, association studies, and sequencing analysis, many of the genes associated with myopia have been identified.<sup>23</sup> Prevalence of myopia has proven to be significantly linked to genetics<sup>24</sup>, and if conclusive findings are made from this study, further analysis of DNA collected from saliva could provide valuable information for posterity. Participants will be asked to spit 2-3 mL of saliva into a self-collection container provided by the study. A slight dryness in the mouth may occur; this will be a one-time collection. Collected saliva samples are for DNA extraction for the DNA to be banked for future, unspecified use. All future research accessing the samples or genetic datasets would be IRB approved and reviewed by the study team on a case-by-case basis.

Participants will be informed that they are donating genetic material, and the most likely outcome is that they will receive no further information regarding those samples.

### 218 1.8 Study Objective

- 219 The purpose of this short-term, pilot, randomized trial is to investigate the efficacy of violet light
- 220 exposure through the BIOS SkyView Lamps at dawn and dusk versus non-violet light exposure through
- 221 Aooshine Bedside Lamps in slowing the progression of myopia in school aged children as an alternative
- 222 to current clinical treatments to determine whether to proceed to a full-scale longer-term randomized
- 223 trial. This decision will be based primarily on assessing responses to light exposure by comparing
- treatment groups on the following outcomes:
- Axial length elongation
- Spherical refractive error
- Quality of life
- The proportion of participants reporting adverse effects
- The proportion of participants reporting >75% light exposure compliance

### 230 1.9 Timing of Intervention and Outcome for Proposed Study

- To evaluate the response to violet light exposure for at least one hour at dawn and at least one hour at
- 232 dusk compared to non-violet light exposure for at least one hour at dawn and at least one hour at dusk,
- this pilot randomized clinical trial (RCT) is proposed. If a reasonable initial response without significant
- adverse effects is found, a subsequent full-scale RCT would further evaluate the effectiveness of violet
- 235 light exposure via the SkyView lamp for myopia treatment. We will define success as violet light
- 236 exposure intervention demonstrating at least 80% non-inferiority compared to the control group.

### 237 **2. Considerations**

### 238 **2.1 Risks**

- 239 Safety testing of both the BIOS SkyView lamp and the Aooshine Bedside Lamp was completed via
- 240 Underwriter Laboratories. (Document: QOVZ.E516890). Both the SkyView lamp (assessment ID: 109744)
- and the Aooshine Bedisde Lamp (assessment ID: 133975) have both been approved for IRB study use by
- 242 CCHMC.
- 243 There is a risk associated with wearing CR-39 lenses, as they are not as impact resistant as polycarbonate
- 244 (mechanical strength class S vs F, respectively). Parents and participants will be educated on the risk via
- the consent form and encouraged to either remove eyeglasses or wear different eyeglasses for activities
- 246 where there is a strong risk of impact to eyeglass lenses (i.e. sports). If participants are assigned to study
- group 2 (CR-39 lenses throughout the day), parents and participants will be reminded verbally of this risk
- using the language present in the consent form.

#### 2.2 Risk of Examination Procedures

- The procedures in this study are part of daily eye care practice in the United States and pose no known
- 251 risks.

249

### 252 2.3 Risk Assessment

- 253 It is the investigator's opinion that the protocol's level of risk falls under DHHS 46.404, which is research
- not involving greater than minimal risk.

256

259

268

269

270

271

272

273

277

278

### 2.4 Reporting of Adverse Events

- There are no expected long-term adverse events associated with violet light exposure. The investigator
- 258 will abide by CCHMC IRB reporting requirements.

### 2.5 Study Costs

- This study will be funded internally through CCHMC RIP grant. The department of ophthalmology will be the final dispenser of funds.
- The subject or his/her insurance provider will be responsible for the costs that are considered standard of care. Because the treatment used in the study is not standard of care, the Enrollment/Randomization,
- 264 Equipment Pickupand 2 Follow-Up visits will be paid for by the study. The cost of the SkyView/Aooshine
- lamp will also be paid for by the study. For subjects who wear prescription lenses and are assigned to a
- 266 group that requires CR-39 or polycarbonate lenses to be worn, the study will provide spectacles and
- lenses from Zenni Optical not to exceed \$80 subject to the following:
  - If the patient/parent desires more expensive frames, they will be responsible for costs that exceed \$80.
  - Lens add-ons and upgrades are at study participant's own expense (e.g., transition lenses, premium polycarbonate lenses).

## 3. Study Outline

| | Enrollment/Randomization | Visit 2: Equipment Recieval | 6-Month Visit | 12- Month Visit |
|---|---|---|---|---|
| | Day ≤0 | Week 4 ± 2 weeks | 6 Months ± 2 weeks | 12 Months ± 2 weeks |
| Informed Consent | X | | | |
| Demographics | X | | | |
| Medical History | х | | X | X |
| Standard Refraction | X | | X | X |
| Cycloplegic Autorefraction | х | | X | X |
| Distance Visual Acuity Testing | x | | X | X |
| Binocular Near Visual Acuity | X | | X | X |
| Monocular Amplitude of Accomodation | X | | X | X |
| Axial Length Measurement | X* | X* | | X** |
| OCTA | X* | X* | | X** |
| Prescribe Refractive Correction If Needed | X | | X | |
| Randomization | х | | | |
| Receive Lamp | | X | | |
| Receive Glasses | | X | | |
| Receive HOBO Sensor | | X | | |
| Receive Automated Wall Plug-In | | X | | |
| HOBO Sensor Data Collection | | | X | X |

274 \*Only required if not able to complete at Enrollment/Randomization Visit.

\*\* Testing may occur at a separate testing visit if testing equipment is unavailable at the 12-Month Visit. This must
occur ± 2 weeks of the 12- Month Visit.

### 4. Enrollment

### 4.1 Eligibility Assessment

- 279 A child is considered for the study after undergoing a routine eye examination (as part of standard care)
- where myopia is identified, and the child appears to meet the eligibility criteria for enrollment. The
- study will be discussed with the child's guardian(s). Guardians who express an interest in the study will
- be given a copy of the informed consent form to read. Written informed consent must be obtained from
- the guardians prior to performing any study-specific procedures that are not part of routine care.
- Participants aged 5 to <13 years with myopia who meet all eligibility criteria will be enrolled in the study.
- Up to 72 participants will be enrolled and randomized in the study.

#### 286 **4.2 Inclusion Criteria**

- Diagnosis of myopia (ICD-10-CM Diagnosis Code H52.13)
- Refractive error meeting the following by cycloplegic autorefraction:
- Myopia -1.00D to -6.00D spherical equivalent (SE) in both eyes
- Astigmatism <= 1.50D in both eyes
- Anisometropia < 1.00D SE
- Complete eye exam with cycloplegic refraction within the past 12 months
- 293 5 to < 13 years of age
- Parent understands the protocol and is willing to accept randomization to 380 nm light or control.
- Parent has a phone (or access to phone) and is willing to be contacted by Investigator's site staff.
- Relocation outside of the area of CCHMC site within the next 12 months is not anticipated.

### 297 **4.3 Exclusion Criteria**

- Current or previous myopia treatment with atropine, pirenzepine or other antimuscarinic agent.
- Current or previous use of bifocals, progressive-addition lenses, or multi-focal contact lenses.
- Current or previous use of orthoK, rigid gas permeable, or other contact lenses being used to reduce myopia progression.
- Current or prior history of manifest strabismus, amblyopia, or nystagmus.
- Abnormality of cornea, lens, central retina, iris, or ciliary body.
- Prior eyelid, strabismus, intraocular, or refractive surgery.
- Down syndrome or cerebral palsy.

### **4.4 Sample Size**

- 307 Up to 72 participants will be enrolled in this study. Up to 24 will be enrolled into the three experimental groups:
- Violet light experimental group with polycarbonate glasses

- Violet light experimental group with CR-39 glasses
- Non-violet control group with CR-39 glasses.

### 312 4.5 Historical Information

- 313 Historical information elicited will include the following: date of birth, sex, race, ethnicity, current
- refractive correction, iris color (brown or not brown), parental history of myopia (0, 1, or 2 parents),
- 315 current medication use, history of and current medical conditions, and myopia treatment history.

### 316 4.6 Survey to Determine Lighting Schedule

- 317 To determine suitable dawn and dusk times for each participant, participants will be asked when they
- 318 typically wake up, eat dinner, and sleep. Additionally, participants will be asked to detail their typical
- evening schedule and any activities that may negatively affect compliance.

### 4.7 Testing at the Enrollment/Randomization Visit

- 321 Testing at the enrollment/randomization visit will include the following:
- 322Standard Refraction

320

- The investigator may use his/her standard refraction technique (with or without cycloplegia) at any
- time during the visit to ensure that the participant meets eligibility criteria with respect to refractive
- 325 correction as described in section 2.5.
- 326 2. Cycloplegic Autorefraction
- 327 Combination Drops (tropicamide 1%, cyclopentolate 1%, phenylephrine 2.5%) one drop twice to
- each eye with 5 minutes between drops. The use of proparacaine prior to the cycloplegic drops is at
- 329 investigator discretion. For each eye, three autorefraction measurements will be taken. For each
- 330 measurement, the autorefractor will yield a final reading (either an individual reading or the
- 331 mean/median of several individual readings, depending on the autorefractor) consisting of sphere,
- 332 cylinder, and axis (see manual of procedures). Each final reading will be converted to a spherical
- equivalent refractive error (SER) and the mean of the 3 SER values for each eye will be used for
- confirming eligibility. A specific autorefractor model is not required for the study; however, each
- participant should have their autorefraction assessed using the same instrument during the entire
- 336 study. The cycloplegic autorefraction should occur at 30 minutes ± 5 minutes from the time the
- second drop was instilled. If eyes are not sufficiently dilated/cyclopleged and/or if the
- dilation/cycloplegia has worn off before all cycloplegic procedures have been performed, another
- drop may be administered, followed by an additional 30-minute wait before testing. The use of
- proparacaine prior to this cycloplegic drop is at investigator discretion.
- 3. Axial Length Measurement and Additional Biometry
- Axial length will be measured 3 times in each eye using optical biometry (e.g., IOLMaster, LENSTAR).
- The following will also be measured 3 times in each eye using optical biometry (e.g., IOLMaster,
- 344 LENSTAR) at the same time as axial length.
- Mean corneal radius (mm to 100th)

346 Anterior chamber depth (mm to 100th) 347 Lens thickness, if available (mm to 100th) 348 A specific instrument is not required for the study; however, each participant should have axial 349 length and additional biometry assessments made using the same instrument during the entire 350 study. 351 If the Enrollment Visit occurs at a time or location that the IOLMaster or LENSTAR is unavailable, the 352 Axial length measurement may be completed at the Equipment Pickup Visit. 353 4. Optical Coherence Tomography Angiography (OCTA) 354 OCTA will be utilized to image retinal vasculature. 3 x 3 mm OCT angiograms will be obtained for 355 each eye. 356 OCTA will be performed using the Heidelberg HRA2 Spectralis device (Heidelberg Engineering, 357 Germany). Using a standardized scanning protocol of 15 degree field of view, 4.4 × 2.9-mm X by Y 358 dimension on the retina, 256 B-scans (12 µm between B-scans), a Z-dimension of 1.9 mm (496 pixels 359 approximated to 3.87  $\mu$ m/pixel), and automatic real-time tracking (ART) of 5; patients will be imaged 360 with macular area OCTA images of superficial vascular complex, deep vascular complex, 361 choriocapillaris and choroid, centered at the fovea. 362 If the Enrollment Visit occurs at a time or location that the Heidelberg HRA2 Spectralis Device is 363 unavailable, the OCTA may be completed at the Equipment Pickup Visit. 4.8 Refractive Correction 364 365 To be eligible for randomization, the participant must be wearing refractive correction in each eye 366 (single vision eyeglasses or soft, daily wear single vision contact lenses with any necessary 367 adjustment for contact lens rotation and vertex distance) that meets the following criteria: 368 1. Myopia (by spherical equivalent) in both eyes must be corrected to within ±0.50 D the 369 investigator's cycloplegic measurement of refractive error. 370 2. Cylinder power in both eyes must be within ±0.50 D of the investigator's standard refraction 371 technique, which can be based on a cycloplegic or non-cycloplegic refraction. 372 3. Cylinder axis for both eyes must be within ±5 degrees of the axis found on the investigator's 373 standard refraction when cylinder power is >= 1.00 D or within ±15 degrees when the cylinder 374 power is < 1.00 D. 375 Measurement of refractive error for assessing the above criteria may be performed as an over 376 refraction or without refractive correction. If the participant meets all eligibility criteria, but their 377 current correction does not meet the requirements for randomization, then new refractive 378 correction (or a change in refractive correction) can be prescribed to meet the requirements. A new 379 (or change) in refractive correction can also be prescribed if the investigator elects to change a

Version 6.0 July 2, 2023

smaller amount of refractive error, but the resulting prescription must meet the criteria above. The

prescribed correction can be single vision eyeglasses or contact lenses. Single vision lenses will be

380

382 paid for by the study; contact lenses will be at the participants' own expense. A pair of eyeglasses is 383 recommended for all participants and may be ordered through Zenni by the study team. 5. Randomization 384 385 **5.1 Randomization Process** 386 Participants eligible for randomization will be randomly assigned in a 1:1:1 distribution respectively to: 387 Violet light experimental group (BIOS SkyView Lamp) with polycarbonate glasses • Violet light experimental group (BIOS SkyView Lamp) with CR-39 glasses 388 389 Non-violet control group (Aooshine Bedside Lamp) with CR-39 glasses 390 The investigator will construct a separate Master Randomization List using a permuted block design 391 stratified by the treatment group. A participant is considered randomized when REDCap randomization 392 process is completed. 393 The participant, parents, testers, and investigators will be masked to treatment group. If the need arises, 394 the investigator may become unmasked after discussion of a specific case with the study team in 395 response to any adverse events. The study coordinator will remain unmasked to the treatment group in 396 order to facilitate the type of equipment and lenses the participant will need. 6. Equipment Pickup Visit 397 398 **6.1 Prescription Glasses** 399 Participants will come back for their Equipment Pickup Visit once the study team has received the 400 glasses shipment from Zenni. These lenses must be used in conjunction with the lamp, therefore must be 401 picked up alongside the lamp. 402 6.2 Study Lamp 403 Participants will receive their lamp at this visit. Patients were randomized at the 404 enrollment/randomization visit and are prepared to receive their respective lamp. The study coordinator 405 will instruct the participant and guardian on the use and setup of the lamp. The HOBO sensor will be 406 attached to the lamp, and participants and guardians will be instructed on how to remove the sensor 407 from the lamp to bring to follow-up visits. 408 6.3 HOBO Sensor 409 Participants will receive the HOBO sensor attached to their lamp. The sensor will be removable to bring 410 to follow-up visits. Participants and guardians will be instructed how to remove the sensor properly, and 411 how to put it back on the lamp. 412 6.4 Automated Wall Plug-In 413 Participants will receive an outlet timer that will be set to the times the parent or guardian has specified

Version 6.0 July 2, 2023

to be their on (dawn) and off (dusk) times. It will be during these times that the child will be asked to be

415 in the room with the light on for at least one hour at dawn and one hour at dusk. This will allow the lamp 416 to turn on and off automatically during the designated times. 6.5 Testing Not Completed at Enrollment 417 418 Participants that were unable to complete testing at the enrollment visit due to unavailability of 419 equipment may have this testing performed at this visit. 420 Axial length measurement (see 4.7.3) 421 OCTA (see 4.7.4) 7. Follow-Up 422 423 7.1 REDCap Daily Surveys 424 Each day, the parent or guardian of the participant will receive a survey via email with two questions as 425 to what times the lamp was used during the dawn hours and dusk hours that day. Parents and guardians 426 will be reminded of the importance of this survey during telephone calls and follow-up visits. 427 This survey will serve as a second point of compliance data to compare to the data received from the 428 HOBO sensor. 429 7.2 Telephone Calls 430 Telephone calls will be made by the study coordinators to the participants and guardians at 2 weeks (+ 3 431 days), 3 months (± 1 month), and 9 months (± 1 month) post Equipment Pickup visit. 432 Coordinators will contact parents to confirm that the BIOS SkyView/Aooshine lamp is working properly, 433 encourage compliance, and question the parent as to whether the child is experiencing any issues with 434 treatment. 435 Additionally, these calls will help maintain direct contact with the parents of the participants, develop 436 and maintain rapport with the family, and assist with scheduling of study visits if needed. 437 7.3 Follow-Up Visits: 6-Month and 12-Month 438 The following will be performed at Follow-Up Visits and recorded in the Follow-Up Visit CRF via Redcap. 439 Medical History 440 o Includes questioning about the occurrence of adverse effects of treatment. Concomitant 441 medications will be recorded, as well as current eyeglasses or contact lenses correction. 442 Compliance Assessment (HOBO sensor data collection) 443 App data will be reviewed and assessments of compliance will be recorded on the 444 Follow-up Examination Form. 445 Standard Refraction 446 The investigator may use their standard refraction technique (with or without 447 cycloplegia) at any time during the visit to ensure that refractive correction meets study 448 criteria at each visit.

Version 6.0 July 2, 2023

Cycloplegic Autorefraction

o See 4.7.2

- 451 Binocular Near Visual Acuity 452 Binocular near visual acuity is measured with participant wearing current refractive 453 correction prior to administration of cycloplegia. 454 **Distance Visual Acuity** Monocular distance visual acuity tested at the start of the exam without cycloplegia in 455 456 current correction. 457 Measurement of best corrected visual acuity in each eye by a study certified visual 458 acuity tester using the E-ETDRS testing protocol. 459 If the vision is more than one line (>= 5 letters) worse than baseline, retest using trial 460 frames or phoropter with the most recent subjective refraction. 461 Monocular Amplitude of Accommodation 462 Measured in their current correction without cycloplegia with a study-specified and provided accommodation near-point rule. 463 464 Axial Length Measurement (12-Month Only) 465 o See 4.7.3 466 OCTA- Performed (12-Month Only) 467 See 4.7.4 468 7.4 Management of Refractive Error 469 Spectacle correction must be updated whenever the investigator's standard refraction technique reveals 470 a change in refractive error. A change in refractive error is defined as any of the following amounts: 471 A difference of >0.75D sphere 472 A difference of >0.75D cylinder 473 • A difference of >0.50D in SE anisometropia 474 A difference in axis of 6 degrees or more when the cylinder is  $\geq$ 1.00D. 475 Whether to update the correction for smaller differences in refraction is at investigator discretion. 476 updated, the refractive correction must meet the requirements described in section 4.7. 477 7.5 Non-Randomized Treatment Other than Refractive Correction 478
- Non-randomized treatment for myopia other than changes in refractive error as described above is not permitted during the study. The investigator must call the principal investigator to discuss the case and obtain approval for an exception prior to initiating non-randomized treatment (including OrthoK, rigid gas permeable, and other contact lenses being prescribed for myopia management).

### 7.6 General Considerations

482

- 483 The study is being conducted in compliance with the policies described in the study policies document,
- 484 with the ethical principles that have their origin in the Declaration of Helsinki, with the protocol
- described herein, and with the standards of Good Clinical Practice.
- Data will be directly collected in electronic CRFs, which will be considered the source data.
- 487 A risk-based monitoring approach will be followed, consistent with the FDA "Guidance for Industry
- Oversight of Clinical Investigations a Risk-Based Approach to Monitoring" (August 2013).

### 8. Miscellaneous Considerations

### 8.1 Participant Withdrawals

489

490

- 491 Parents may withdraw their child from the study at any time. If the parents indicate that they want to
- 492 withdraw their child from the study, the investigator should attempt to speak with the parents personally
- 493 to determine the reason. If their interest is in transferring the child's care to another eye care provider,
- every effort should be made to comply with this and at the same time, try to keep the participant in the
- 495 study under the new provider's care.

### 496 **8.2 Discontinuation of Study**

- The study may be discontinued by the study team prior to the pre-planned completion of enrollment
- 498 and follow-up for all participants.

## 499 8.3 Payment to Participants

- 500 The parent/guardian of each participant will be compensated \$50 by ClinCard upon completion of the
- 501 Enrollment/Randomization Visit, Equipment Pickup Visit, 6-Month Visit, and 12-Month Visits, for a
- 502 maximum of \$250.

### **8.4 Costs Covered by the Study**

- The study will pay for the office visits that are part of the study (Enrollment/Randomization Visit,
- 505 Equipment Pickup Visit, 6-Month Visit, and 12-Month Visit).
- 506 The study will pay for the following:
- BIOS SkyView/Aooshine lamp will be provided to each participant at no cost.
- Eyeglasses will be ordered at enrollment (if needed).
- Frames and Lenses will be ordered by the study team from Zenni.
- Lens changes will be provided at 6 months if a change is required, and the lenses will be ordered by the study team through Zenni.

### 512 8.5 Costs Not Covered by the Study

- 513 The study will not pay for eyeglasses obtained elsewhere (the study pays for glasses if needed through
- Zenni only). The study will not pay for contact lenses.

### 9. Data Storage and Analysis

#### 516 **9.1 Analysis**

515

- 517 <u>Primary Analyses</u>
- 518 The primary analysis will be an experimental vs control group comparison of change from baseline to 12
- 519 months in spherical equivalent refractive error (SER), as measured using cycloplegic autorefraction. At
- 520 baseline and all follow-up visits, the mean of the three readings from autorefraction in each eye will be
- 521 calculated and then the mean of both eyes for each participant will be used for the analysis. If fewer
- than 3 readings are available in each eye, the mean of available readings will be used for each eye to
- obtain the mean of both eyes for each participant.

The treatment group difference (violet vs. non-violet light) and a 95% confidence interval will be calculated based on the model estimates at 12 months.

### 526 Secondary Analyses

- Difference in change in axial length at 6 and 12 months between the violet and non-violet light group
  - Compliance will be assessed at each follow up and described as excellent (76%-100%), good (51%-75%), fair (26%-50%) or poor (<25%).

#### 9.2 Decision Guideline

- 532 The data collected in this short-term, pilot randomized clinical trial will primarily be used to determine
- 533 whether to proceed to a full-scale, longer-term randomized trial of violet light vs control non-violet. The
- side effect profiles in the experimental and control groups will also be considered when deciding
- whether to proceed with a full-scale trial.
- 536 The decision guideline for determining whether to proceed to a full-scale randomized trial will be based
- on the primary and secondary outcomes at study conclusion.

### 538 9.3 Data Safety Monitoring Plan

- The participants in this study are patients routinely seen by the investigator or his colleagues as part of
- standard clinical care at CCHMC, Division of Pediatric Ophthalmology. Participants will continue to be
- followed clinically by either the investigator or the referring clinicians in addition to attending the study
- 542 visits.

529

530

531

- During the study, participants are observed closely to detect occurrences of any adverse events or
- complications that may have arisen. At each study visit, the participants and their guardians will be asked
- questions regarding the occurrence of adverse events to determine whether any complications or
- adverse events might have occurred since the previous visit.
- 547 In the case of a suspected adverse event, further testing may be performed, and non-study treatment
- may be initiated to ensure patient safety.

### **9.4 Source Documents and Case Report Forms**

- Adequate records will be maintained for the study including participant medical records, test reports,
- 551 signed informed consent forms, adverse event reports, and information regarding participant
- discontinuation and reasons for discontinuation. All original source documentation will be stored
- 553 electronically in the password-protected CCHMC shared-drive or in a locked filing cabinet located in the
- investigator's office or research coordinator's workspace.
- 555 In accordance with 21 CFR 50, guardians will provide written informed consent for participation in this
- 556 study.

557

#### 9.5 Changes to Protocol

- The investigator will notify the IRB of any unanticipated problem requiring a change in the protocol to
- eliminate apparent immediate hazard to a subject per CCHMC Research Policy, R-18. Changes that affect

| 560<br>561 | the scientific soundness of the study or the rights, safety, or welfare of human subjects will be submitted to the IRB in an amendment prior to implementation. | |
|---|---|---|
| 562 | | |
| 563 | | |
| 564 | | |
| 565 | | |
| 566 | 10. | 10. References |
| 567<br>568 | 1. | Holden, B. A. et al. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. <i>Ophthalmology</i> (2016) doi:10.1016/j.ophtha.2016.01.006. |
| 569<br>570 | 2. | Theophanous, C. et al. Myopia prevalence and risk factors in children. Clin. Ophthalmol. (2018) doi:10.2147/OPTH.S164641. |
| 571 | 3. | Foster, P. J. & Jiang, Y. Epidemiology of myopia. Eye (2014) doi:10.1038/eye.2013.280. |
| 572<br>573<br>574 | 4. | Praveen, M. R., Vasavada, A. R., Jani, U. D., Trivedi, R. H. & Choudhary, P. K. Prevalence of Cataract Type in Relation to Axial Length in Subjects with High Myopia and Emmetropia in an Indian Population. <i>Am. J. Ophthalmol.</i> (2008) doi:10.1016/j.ajo.2007.07.043. |
| 575<br>576<br>577 | 5. | Mitchell, P., Hourihan, F., Sandbach, J. & Wang, J. J. The relationship between glaucoma and myopia: The blue mountains eye study. <i>Ophthalmology</i> (1999) doi:10.1016/S0161-6420(99)90416-5. |
| 578<br>579 | 6. | Risk factors for idiopathic rhegmatogenous retinal detachment. <i>Am. J. Epidemiol.</i> (1993) doi:10.1093/oxfordjournals.aje.a116735. |
| 580<br>581 | 7. | Walline, J. J. Myopia control: A review. <i>Eye and Contact Lens</i> (2016) doi:10.1097/ICL.000000000000000000000000000000000000 |
| 582<br>583 | 8. | Walline, J. & Smith, M. Controlling myopia progression in children and adolescents. <i>Adolesc. Health. Med. Ther.</i> (2015) doi:10.2147/ahmt.s55834. |
| 584<br>585 | 9. | Leo, S. W. et al. Current approaches to myopia control. <i>Current Opinion in Ophthalmology</i> (2017) doi:10.1097/ICU.000000000000367. |
| 586<br>587<br>588 | 10. | Lam, C. S. Y., Tang, W. C., Tse, D. Y. Y., Tang, Y. Y. & To, C. H. Defocus Incorporated Soft Contact (DISC) lens slows myopia progression in Hong Kong Chinese schoolchildren: A 2-year randomised clinical trial. <i>Br. J. Ophthalmol.</i> (2014) doi:10.1136/bjophthalmol-2013-303914. |
| 589<br>590<br>591 | 11. | He, M. et al. Effect of time spent outdoors at school on the development of myopia among children in China a randomized clinical trial. <i>JAMA - J. Am. Med. Assoc.</i> (2015) doi:10.1001/jama.2015.10803. |
| 592<br>593 | 12. | Wu, P. C., Tsai, C. L., Wu, H. L., Yang, Y. H. & Kuo, H. K. Outdoor activity during class recess reduces myopia onset and progression in school children. <i>Ophthalmology</i> (2013) |

| 594 | | doi:10.1016/j.ophtha.2012.11.009. |
|---|---|---|
| 595<br>596 | 13. | Rose, K. A. et al. Myopia, lifestyle, and schooling in students of Chinese ethnicity in Singapore and Sydney. <i>Arch. Ophthalmol.</i> (2008) doi:10.1001/archopht.126.4.527. |
| 597<br>598<br>599 | 14. | Sherwin, J. C. <i>et al.</i> The association between time spent outdoors and myopia in children and adolescents: A systematic review and meta-analysis. <i>Ophthalmology</i> (2012) doi:10.1016/j.ophtha.2012.04.020. |
| 600<br>601 | 15. | Xiong, S. et al. Time spent in outdoor activities in relation to myopia prevention and control: a meta-analysis and systematic review. Acta Ophthalmologica (2017) doi:10.1111/aos.13403. |
| 602<br>603<br>604 | 16. | Jin, J. X. <i>et al.</i> Effect of outdoor activity on myopia onset and progression in school-aged children in northeast china: The sujiatun eye care study. <i>BMC Ophthalmol.</i> (2015) doi:10.1186/s12886-015-0052-9. |
| 605<br>606 | 17. | Torii, H. <i>et al.</i> Violet Light Exposure Can Be a Preventive Strategy Against Myopia Progression. <i>EBioMedicine</i> (2017) doi:10.1016/j.ebiom.2016.12.007. |
| 607<br>608 | 18. | Torii, H., Ohnuma, K., Kurihara, T., Tsubota, K. & Negishi, K. Violet Light Transmission is Related to Myopia Progression in Adult High Myopia. <i>Sci. Rep.</i> (2017) doi:10.1038/s41598-017-09388-7. |
| 609<br>610 | 19. | Nguyen, M. T. T. et al. An opsin 5—dopamine pathway mediates light-dependent vascular development in the eye. <i>Nat. Cell Biol.</i> (2019) doi:10.1038/s41556-019-0301-x. |
| 611<br>612<br>613 | 20. | Zhou, X., Pardue, M. T., Iuvone, P. M. & Qu, J. Dopamine signaling and myopia development: What are the key challenges. <i>Progress in Retinal and Eye Research</i> (2017) doi:10.1016/j.preteyeres.2017.06.003. |
| 614<br>615<br>616 | 21. | Wang, M., Schaeffel, F., Jiang, B. & Feldkaemper, M. Effects of light of different spectral composition on refractive development and retinal dopamine in chicks. <i>Investig. Ophthalmol. Vis. Sci.</i> (2018) doi:10.1167/iovs.18-23880. |
| 617<br>618<br>619 | 22. | Jiang X, Pardue MT, Mori K, Ikeda S, Torii H, D'Souza S, Lang RA, Kurihara T, Tsubota K. "Violet light suppresses lens-induced myopia via neuropsin (OPN5) in mice." <i>Proc Natl Acad Sci.</i> 2020. ( <i>in review</i> ) |
| 620<br>621<br>622 | 23. | Yap M, Wu M, Liu ZM, Lee FL, Wang SH. Role of heredity in the genesis of myopia. Ophthalmic Physiol Opt. 1993;13:316–9. |
| 623<br>624<br>625 | 24. | Ip JM, Huynh SC, Robaei D, Rose KA, Morgan IG, Smith W, Kifley A, Mitchell P. Ethnic Differences in the impact of parental myopia: findings from a population-based study of 12-year-old Australian children. Invest Ophthalmol Vis Sci. 2007;48:2520–8. |
| 626<br>627 | 25. | BIOS. WELL Building Standard: Circadian Lighting Design. Jan 2020. <a href="https://bioslighting.com/human/well-building-standard/">https://bioslighting.com/human/well-building-standard/</a> |
| 628 | 26. | BIOS. SkyView Wellness Table Lamp, Jan 2020, https://bioslighting.com/product/SkyView- |

wellness-table-lamp/